CLINICAL TRIAL: NCT05638204
Title: A Randomized Controlled Study on the Effectiveness of the Suicidal Crisis Intervention (SCI)
Brief Title: Effectiveness of the Suicidal Crisis Intervention (SCI)
Acronym: RCT SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2022-0376
Record Dates: First submitted 2022-11-08; First posted 2022-12-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Suicide; Suicidal Ideation; Suicide, Attempted
MeSH Terms: conditions — Suicide; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial using permuted block randomization with variable block sizes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group received the Suicidal Crisis Intervention( SCI) in addition to their treatment as usual.
  Interventions: Behavioral: Suicidal Crisis Intervention (SCI)
- Control Group (No Intervention): Participants in the control group received their treatment as usual.

INTERVENTIONS:
Behavioral: Suicidal Crisis Intervention (SCI) — This study's experimental condition consisted of the Suicidal Crisis Intervention (SCI), developed by the Flemish Centre of Expertise of Suicide prevention. The SCI aims to provide tools for dealing with future suicidal crises for people after a suicidal crisis or suicide attempt. The intervention attempts to provide insight into the suicidal crisis by giving suicidality meaning within the life history. It aims to increase motivation for specialized care and therefore facilitate continuity of care. In addition, the method also wants to involve the close relative(s) of the suicidal person in the treatment. The SCI offers care providers a clear structure and handles to do this within a short period of time (4 sessions). Within the SCI are a number of crucial elements: the therapeutic relationship, involving loved ones, person-centred care, the Integrated Explanatory Model for Suicidal Behavior (Van Heeringen, 2007), the safety plan (Stanley & Brown, 2012) and continuity of care.
  Arms: Intervention Group

SUMMARY:
The main objective of this project is to be able to offer a new, specific evidence-based short-term treatment method, the Suicidal Crisis Intervention (SCI), to reduce suicidality. In addition, this study aims to investigate the influence of SCI on other important aspects of suicidality (secondary goal) such as hopelessness, defeat, entrapment, and interpersonal needs.

DETAILED DESCRIPTION:
Research has extensively shown that a previous suicide attempt or a history of suicide attempts are important predictors of suicide death. It is therefore important to provide people with appropriate care after a suicide attempt to limit this risk.

Although this risk factor (previous attempts) is known, the number of interventions developed for this risk group is limited.

Based on these findings, a short-term treatment trajectory was developed for people after a suicide attempt or a suicidal crisis in Flanders, called the Suicidal Crisis Intervention (SCI). This was inspired by the ASSIP treatment trajectory and the safety plan was also given a significant place within the treatment. In addition, the importance of relatives and social support is emphasized by involving relatives in this treatment. Throughout this treatment, further (treatment) goals are drawn up, in order to generate hope for improvement and to facilitate continuity of care. More information about the concrete content of SCI will follow later in this protocol. A pilot study is currently being conducted to assess the feasibility of this treatment, as well as the experience of patients, relatives and care providers. Based on this, the SCI will be further updated for this effectiveness study.

There are currently no specific evidence-based short-term treatment methods in Flanders for people after a suicidal crisis or suicide attempt. The primary research question is therefore: 'Is the Suicidal Crisis Intervention (SCI) in Flanders an effective short-term treatment method for people after a suicidal crisis or suicide attempt?'.

The main objective of this project is to be able to offer a new, specific short-term treatment method that has been scientifically proven to reduce suicidality. In addition, we want to investigate the influence of SCI on other important aspects of suicidality (secondary goal) such as hopelessness, defeat, entrapment, and interpersonal needs.

ELIGIBILITY:
Inclusion Criteria Patient:

* After a suicide attempt or suicidal crisis
* ≥ 18 years
* Availability of a smartphone, tablet and/or computer with internet access,
* Dutch-speaking.

Exclusion Criteria Patient:

* Limited comprehension, cognitive impairment
* Psychotic disorder
* Unsuitable for individual therapy
* Receiving other forms of care is not an exclusion criterion.

Inclusion Criteria Close one:

* close one of the patient
* ≥ 18 years
* Dutch- speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in suicidality: Beck Scale for Suicide Ideation (BSI; Beck & Steer, 1991) | Change in baseline to post-test [42 days after randomization], to follow-up 1 [132 days after randomization] and to follow-up 2 [222days after randomization]
  The BSI is a 21-item self-report questionnaire. Each item is rated on a scale from 0 to 2, resulting in a total score ranging from 0 to 38.

SECONDARY OUTCOMES:
Change in suicidal behaviour | Change in baseline to post-test [42 days after randomization], to follow-up 1 [132 days after randomization] and to follow-up 2 [222days after randomization]
  Using two questions participants will be asked whether they have experienced suicidal thoughts (lifetime and since last measure, or last year for baseline) and whether they attempted suicide (lifetime and since last measure, or last year for baseline)
Change in hopelessness: The Beck Hopelessness Scale (BHS; Beck et al., 1974) | Change in baseline to post-test [42 days after randomization], to follow-up 1 [132 days after randomization] and to follow-up 2 [222days after randomization]
  A 20-item self-report questionnaire to measure hopelessness in adolescents and adults. Each item is rated as 'true' (score = 1) or 'false' (score = 0) for them over the past week, resulting in a total score ranging from 0 to 20, with higher scores indicating higher levels of hopelessness (worse outcome).
Change in defeat: Defeat Scale (DS; Gilbert & Allen, 1998; Griffiths et al., 2015) - short version | Change in baseline to post-test [42 days after randomization], to follow-up 1 [132 days after randomization] and to follow-up 2 [222days after randomization]
  A 4-item self-report questionnaire to measure defeat on a five-point Likert scale. A total score ranging from 0 to 16 is obtained, with higher scores indicating more perceptions of defeat (worse outcome).
Change in entrapment: Entrapment Scale (ES; Gilbert & Allen, 1998; Griffiths et al., 2015) - short version | Change in baseline to post-test [42 days after randomization], to follow-up 1 [132 days after randomization] and to follow-up 2 [222days after randomization]
  A 4-item self-report questionnaire to measure entrapment on a five-point Likert scale. A total score ranging from 0 to 16 is obtained, with higher scores indicating more perceptions of entrapment (worse outcome).
Change in isolation: Interpersonal Needs Questionnaire (INQ; Van Orden et al., 2012; Hill et al., 2015) - short version | Change in baseline to post-test [42 days after randomization], to follow-up 1 [132 days after randomization] and to follow-up 2 [222days after randomization]
  This is a 10-item questionnaire where each item is rated on a 7-point Likert scale with 1= Not at all true for me, 4 = somewhat true for me and 7 = very true for me.
Change in (prepared to follow) follow-up care [own questionnaire] | Change in baseline to post-test [42 days after randomization], to follow-up 1 [132 days after randomization] and to follow-up 2 [222days after randomization]
  To assess whether participants receive follow-up care or are prepared to receive follow-up care, 14 questions were asked. About which psychological [none, GP, psychologist, psychiatrist, other health care worker, residential care, waiting list], medical [no medication, pain killers, tranquilizers/anxiolytics, sleeping pills, antidepressants, antipsychotics, other] treatment they were currently receiving, they started/stopped/changed since the start of the study and or prepared to receive. This will not result in a total score, but instead will be used as a descriptive questionnaire.
Treatment satisfaction [own questionnaire] | Post-test [42 days after randomization]
  To investigate how patients of the intervention group experienced the SCI, some evaluative questions are asked. Participants are asked to indicate how many sessions they received, how they would rate the treatment [0-10], what they thought of the number and length of sessions [too little/short, good, too many/long], rate to what degree they agreed [strongly disagree, disagree, neutral, agree, strongly agree, not applicable] with 8 statements about the treatment, and 2 open questions about the strengths, weaknesses of the treatment.

OTHER OUTCOMES:
Treatment evaluation by close one [own questionnaire] | Post-test [42 days after randomization]
  To investigate how close ones of the patients in the intervention group experienced the SCI, some evaluative questions are asked. Participants are asked to indicate how many sessions they received, how they would rate the treatment [0-10], what they thought of the number and length of sessions [too little/short, good, too many/long], rate to what degree they agreed [strongly disagree, disagree, neutral, agree, strongly agree, not applicable] with 8 statements about the treatment, and 2 open questions about the strengths, weaknesses of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, Phd, Principal Investigator — University Ghent
Locations (12):
- Belgium (12):
  - Psychiatrisch Centrum Sint Amandus (incl. Mobiel Crisis Team), Beernem
  - Medisch Centrum St. Jozef, Bilzen
  - Mobiel Crisis Team zorggroep Multiversum, Boechout
  - Openbaar Psychiatrisch Zorgcentrum Geel, Geel
  - UZ Gent, Ghent
  - AZ Groeninge (incl. Mobiel Crisis Team Kortrijk), Kortrijk
  - Psychiatrisch Ziekenhuis Heilige Familie Kortrijk, Kortrijk
  - Psychiatrisch Centrum Ariadne, Lede
  - Openbaar Psychiatrisch Zorgcentrum Rekem, Rekem
  - Algemeen Ziekenhuis Glorieux, Ronse
  - Psychiatrisch Ziekenhuis Sint Lucia (incl. Mobiel Team Acute Zorgen), Sint-Niklaas
  - Bethanië GGZ (incl. mobiel crisis team SARA Het Veer), Zoersel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris EC, Barraclough B. Suicide as an outcome for mental disorders. A meta-analysis. Br J Psychiatry. 1997 Mar;170:205-28. doi: 10.1192/bjp.170.3.205. PMID 9229027
- [Background] Hawton K, Zahl D, Weatherall R. Suicide following deliberate self-harm: long-term follow-up of patients who presented to a general hospital. Br J Psychiatry. 2003 Jun;182:537-42. doi: 10.1192/bjp.182.6.537. PMID 12777346
- [Background] Nordentoft M. Crucial elements in suicide prevention strategies. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Jun 1;35(4):848-53. doi: 10.1016/j.pnpbp.2010.11.038. Epub 2010 Dec 2. PMID 21130823
- [Background] Michel, K., & Gysin-Maillart, A. (2015). ASSIP - Attempted Suicide Short Intervention Program: A manual for clinicians. Hogrefe Publishing.

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT05638204/SAP_000.pdf